CLINICAL TRIAL: NCT06005168
Title: Comparison of a Morphomic-Based to the Standard-of-Care-Based Cefazolin Dose for Antimicrobial Prophylaxis
Acronym: MorphAbxPKSurg
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Manjunath Prakash Pai, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00222771; R01HS027183 (AHRQ)
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Surgical Prophylaxis
Keywords: Surgical Prophylaxis; Pharmacokinetics; Cefazolin; Obesity; Morphomics; Colorectal
MeSH Terms: conditions — Obesity | interventions — Cefazolin; Injections

STUDY DESIGN:
Intervention Model Description: The current model for dosing the drug cefazolin includes the selection of 2 grams if the individual weighs less than 120 kg and 3 grams if they weigh 120 kg or more. The morphomic-based model defined the choice of 2 grams versus 3 grams of cefazolin based on kidney function and body depth.
Masking Description: This is open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (No Intervention): The patients assigned to this group have cefazolin dose assignments based on body weight, which is the standard of care.
- Morphomic-based (Active Comparator): The patients assigned to this group have cefazolin dose assignments based on body depth and kidney function.
  Interventions: Drug: Cefazolin for Injection

INTERVENTIONS:
Drug: Cefazolin for Injection — 2 grams or 3 grams based on standard of care or morphomic-based decision
  Arms: Morphomic-based

SUMMARY:
The goal of this clinical study is to compare the dosing of an antibiotic in overweight patients having surgery. The main question[s] it aims to answer are:

* Are the antibiotic concentrations in blood and fat tissue in patients that are overweight sufficient to prevent the chance of infection?
* Can dosing using body composition rather than body weight improve the chance of achieving good antibiotic concentrations in overweight patients? Participants will allow us to collect small amounts of blood and fat tissue during their regularly scheduled surgery.

Researchers will compare differences in antibiotic concentrations based on dosing by standard of care (body weight based) versus body composition.

DETAILED DESCRIPTION:
The risk of surgical site infections are higher in patients with obesity compared to non-obese adults. Our group has previously demonstrated that radiologic measures of abdominal subcutaneous fat are associated with surgical site infection risk in patients undergoing colorectal surgeries, which could reflect suboptimal antibiotic exposure in these patients. Therefore, we hypothesized that measures of abdominal size and composition in patients undergoing colorectal surgery would be more predictive of antimicrobial pharmacokinetics in this tissue compartment than the current standards of body weight and BMI. We confirmed this hypothesis and identified kidney function and body depth (by morphomics) to be predictive of cefazolin exposure in target tissue. Morphomics is a technology that transforms existing computed tomography data into body measures and composition. This study is a head-to-head comparison of this new proposed morphomic test regimen to the standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Accessible abdominal computed tomography scan prior to surgery
2. Adult patients > 18 years of age
3. Body Mass Index ≥ 25 kg/m^2
4. Expected to receive cefazolin prior to surgical incision
5. Estimated creatinine clearance ≥90 mL/min

Exclusion Criteria:

1. History of a hypersensitivity reaction to penicillin or cephalosporin
2. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Proportion of Concentration Target Attainment | 4 hours
  Proportion of patients achieving at least 3.2 hours of time above 2 mcg/mL (MIC90) in subcutaneous fat tissue with the standard of care compared to morphomic-based dosing

SECONDARY OUTCOMES:
Cefazolin exposure based on body depth | 4 hours
  Compare the area under the curve from time 0 to 4 hours (AUC0-4) in plasma and subcutaneous fat in patients with a body depth above and below 350 mm
Cefazolin exposure based on kidney function | 4 hours
  Compare the area under the curve from time 0 to 4 hours (AUC0-4) in plasma and subcutaneous fat in patients with an estimated creatinine clearance above and below 120 mL/min

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No